CLINICAL TRIAL: NCT07005557
Title: Study Evaluating Node-positive, ER+/HER2- In Older (≥65 Years) Breast Cancer Patients for Chemotherapy Exemption: A Randomized, Open-label, Multicenter Phase III Clinical Trial
Brief Title: Chemo-free in Older (≥65) Node-Positive ER+/HER2- Breast Cancer
Acronym: SENIOR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N089
Record Dates: First submitted 2025-05-03; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Adjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Chemotherapy, endocrine therapy, or CDK4/6 inhibitors, administered at the physician's discretion.
  Interventions: Drug: Chemotherapy; Drug: CDK4/6 Inhibitor; Drug: Endocrine therapy
- Chemo-free (Experimental): A chemotherapy-sparing approach using CDK4/6 inhibitor combined with aromatase inhibitor (minimum 5-year duration).
  Interventions: Drug: CDK4/6 Inhibitor; Drug: Endocrine therapy

INTERVENTIONS:
Drug: Chemotherapy — Chemotherapy options at physician's discretion: TC, EC-T(wP), or capecitabine.
  Arms: Control
Drug: CDK4/6 Inhibitor — All patients will receive CDK4/6 inhibitor (abemaciclib/ribociclib/dalpiciclib/palbociclib)
Drug: Endocrine therapy — Endocrine therapy (letrozole/anastrozole/exemestane)

SUMMARY:
This study is a prospective, open-label, multicenter, randomized controlled Phase III clinical trial. Based on the use of CDK4/6 inhibitors in endocrine-sensitive luminal-type (ER+/HER2-) breast cancer, it aims to explore the possibility of chemotherapy exemption in elderly patients (aged >65 years) with lymph node-positive, HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

-1. Age: Female patients aged ≥65 years. 2. Disease Status: Histologically confirmed early-stage breast cancer after surgery with ER expression ≥50% AND one of the following:

1. ≥4 positive lymph nodes
2. 1-3 positive lymph nodes plus at least one of the following high-risk features: i. High-risk multigene assay result ii. Primary tumor size >2 cm iii. Histologic grade 3 iv. Lymphovascular invasion (LVI) positive v. Ki-67 >20% 3. Treatment Acceptance: Willing to receive adjuvant CDK4/6 inhibitor therapy. 4. Performance Status: ECOG score 0-2. 5. Adequate Organ Function:

a) Hematology (within 14 days, no transfusion): i. Hemoglobin (Hb) ≥90 g/L ii. Absolute neutrophil count (ANC) ≥1.5×10⁹/L iii. Platelets (PLT) ≥100×10⁹/L b) Biochemistry: i. Total bilirubin (TBIL) ≤1.5×ULN ii. ALT/AST ≤3×ULN iii. Serum creatinine (Cr) ≤1×ULN iv. Estimated creatinine clearance (CrCl) >50 mL/min (Cockcroft-Gault formula) 6. Consent & Compliance: Willing to participate, sign informed consent, and comply with follow-up.

Exclusion Criteria:

* 1. Patients who have received neoadjuvant therapy (including chemotherapy, targeted therapy, radiotherapy, or endocrine therapy).

  2. Bilateral breast cancer. 3. History of other malignancies, except: Cured basal cell carcinoma of the skin； Carcinoma in situ of the cervix 4. Distant metastasis (any site). 5. Any T4 lesion (UICC 1987 TNM staging), including: Skin invasion; Fixed mass adherence; Inflammatory breast cancer 6. Concurrent participation in other clinical trials. 7. Severe organ dysfunction (cardiac, pulmonary, hepatic, or renal), including:

  a) LVEF <50% (by echocardiography) b) Major cardiovascular/cerebrovascular events within 6 months before randomization: i. Unstable angina ii. Chronic heart failure iii. Uncontrolled hypertension (>150/90 mmHg) iv. Myocardial infarction or stroke c) Poorly controlled diabetes mellitus d) Severe hypertension 8. Known allergy to taxane-based drugs or their excipients. 9. Severe or uncontrolled infections. 10. History of psychoactive drug abuse (unable to abstain) or psychiatric disorders.

  11. Patients deemed ineligible by investigator assessment. 12. Refusal to receive adjuvant CDK4/6 inhibitor therapy.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1244 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2030-05-15 (Estimated); Study Completion 2035-05-15 (Estimated)

PRIMARY OUTCOMES:
5-years Invasive disease free survival | 5 years
  5-year invasive disease-free survival (iDFS), defined as the time from randomization to the first occurrence of: local recurrence, distant metastasis, contralateral invasive breast cancer, death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 5 years
  OS is defined as the time from randomisation until the date of death due to any cause.
Safety including adverse events (AEs), severe adverse events (SAEs) and adverse events of special interest (AESI). | Up to approximately 3 years
  Incidence of AEs, SAE, AESIs (interstitial lung disease, LVEF decrease), AEs resulting in study intervention interruption and discontinuation, etc.
Geriatric assessment (G-8) | Up to approximately 3 years
  • Modified Geriatric-8 (G-8) screening tool
Clinical Frailty Scale | Up to approximately 3 years
  Clinical Frailty Scale (CFS, version 2.0)

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Shao, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No